CLINICAL TRIAL: NCT06222918
Title: Investigation of the Effect of Deep Margin Elevation Technique on the Clinical Performance of Endocrown Restorations Produced by Computer-Aided Design and Computer-Aided Manufacturing (CAD/CAM) System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Onur Adson, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22110
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Dental Caries
Keywords: CAD/CAM; Endocrown; Deep Margin Elevation; İndirect
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supragingival margins (No Intervention)
- Subgingival margins (G-ænial Universal Injectable) (Active Comparator): Matrix: Methacrylate monomer %31. Fillers: Silica, Barium Glass %69
  G-ænial Universal injectable is a light-cured, radiopaque universal high-strength composite that can be used for all restorative indications while offering excellent viscosity and perfect direct syringe application. It has enhanced thixotropic properties that allow you to create the most beautiful & durable restorations with a minimum of manipulation.
  Interventions: Procedure: Deep Margin Elevation (G-ænial Universal Injectable)

INTERVENTIONS:
Procedure: Deep Margin Elevation (G-ænial Universal Injectable) — Deep margin elevation (DME), or coronal margin relocation (CMR), is a procedure used to raise or reposition sub-gingival margins into supra-gingival margins using several materials to increase marginal integrity and bonding strength
  Arms: Subgingival margins (G-ænial Universal Injectable)

SUMMARY:
The aim of this clinical study is to investigate the impact of the deep margin elevation technique on the clinical performance of CAD/CAM endocrown restorations in deep Class II cavities.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of the deep margin elevation technique on the clinical performance of endocrown restorations made from nano-ceramic blocks produced using the CAD/CAM system for class II cavities with deep margins. Factors such as color harmony with adjacent teeth and restorations, discoloration, anatomical form continuity, adaptation, secondary caries, and retention will be examined in the nano-ceramic block material.

Various treatment options are available for the restoration of posterior group teeth. Factors such as restoration material, condition of supporting tooth tissue, patient habits, and clinical protocols affect the lifespan of restorations. Advances in tooth preparations ensure the preservation of sound tooth structure and the longevity of restorations.

The CAD/CAM system is a technology used in dentistry, consisting of three essential elements: data acquisition, design, and production. With this system, dentists can design and produce restorations such as veneers, crowns, and bridges using digital modeling and manufacturing methods.

The restoration of endodontically treated teeth may require different approaches than post-core and crown restorations that can affect mechanical resistance. The development of adhesive techniques and the importance of minimally invasive dentistry have led to new therapeutic approaches, such as monolithic endocrown restorations fixed to the pulp chamber and cavity margins.

Dental adhesion is the attractive force between the tooth surface and the applied material, and dentin bonding systems have been developed to ensure adhesion between the two structures. These systems enhance adhesion by increasing dentin surface energy and facilitating the spread of adhesive resin into the dentin.

Procedures such as isolation, measurement, cementation, and residual cement cleaning can be challenging in cases with deep margins. Clinical strategies can assist in overcoming isolation difficulties in subgingival margin areas where adhesive procedures are applied.

The restoration of teeth with advanced substance loss can be a challenging process for operators, and the selection of the correct treatment plan is crucial. This clinical research aims to examine the impact of the deep marginal elevation technique on the clinical performance of CAD/CAM-produced endocrown restorations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without any uncontrolled systemic diseases.
* Individuals aged between 18 and 65 years.
* Individuals who pay attention to oral hygiene by brushing their teeth twice a day.
* Patients with at least one canal-treated posterior tooth, multiple cusp loss, and at least one tooth wall loss identified during intraoral examination.
* Patients who have successfully completed periodontal and endodontic treatments and do not exhibit any subjective symptoms.

Voluntary individuals who agree to participate in the study and sign the informed consent form will be included in the research.

Exclusion Criteria:

* Individuals with uncontrolled systemic diseases.
* Individuals with mental retardation who cannot establish cooperation.
* Individuals with advanced periodontal disease.
* Individuals using removable partial dentures.
* Individuals with bruxism.
* Individuals with malocclusion.
* Patients with advanced substance loss requiring extraction of the relevant tooth, and individuals with deep margins requiring periodontal interventions.

Individuals who, after being informed about the study, choose not to read the informed consent form and decline to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2024-04-25 (Estimated)

PRIMARY OUTCOMES:
Retention | From baseline to 24 month
  Observers evaluated the restorations was performed using the United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No loss of restorations materyal. Charlie: Any loss of restorative material
Marginal discoloration | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding Marginal staining. Marginal staining was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scorsese: Alfa: No discoloration. Bravo: Discoloration without. Charlie:Discoloration with penetration in pulpal direction
Marginal Adaptation | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; Alfa: Closely adapted, no visible crevice. Bravo: Visible crevice, explorer will penetrate. Charlie: Crevice in which dentin is exposed
Seconder Caries | From baseline to 24 month
  Observers evaluated the restorations was performed using the United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No caries presented. Charlie Caries present

CONTACTS AND LOCATIONS:
Overall Officials: Şükran Bolay, Prof., Principal Investigator — Hacettepe University; Taha Yasin Sarıkaya, Principal Investigator — Hacettepe University; Onur Adson, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Veneziani M. Adhesive restorations in the posterior area with subgingival cervical margins: new classification and differentiated treatment approach. Eur J Esthet Dent. 2010 Spring;5(1):50-76. PMID 20305873
- [Background] Juloski J, Koken S, Ferrari M. Cervical margin relocation in indirect adhesive restorations: A literature review. J Prosthodont Res. 2018 Jul;62(3):273-280. doi: 10.1016/j.jpor.2017.09.005. Epub 2017 Nov 15. PMID 29153552
- See also: Related İnfo — https://www.gc.dental/europe/en/products/gaenialuniversalinjectable